CLINICAL TRIAL: NCT02871960
Title: Evaluation of Surgical Stress and Immune Response After Minimally Invasive Colorectal Surgery (ESSIMIC)
Brief Title: Surgical Stress and Colorectal Surgery
Acronym: ESSIMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Milone, Professor of Surgery, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoboticUnina2016
Record Dates: First submitted 2016-07-21; First posted 2016-08-18 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2019-12

CONDITIONS: Surgical Stress and Immune Function
MeSH Terms: interventions — Robotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic colectomy (Experimental): Patients undergoing robotic colectomy for colorectal cancer
  Interventions: Procedure: Robotic and Laparoscopic Colectomy
- Laparoscopic colectomy (Active Comparator): Patients undergoing laparoscopic colectomy for colorectal cancer
  Interventions: Procedure: Robotic and Laparoscopic Colectomy

INTERVENTIONS:
Procedure: Robotic and Laparoscopic Colectomy

SUMMARY:
The purpose of this study is to evaluate surgical stress and immune function after robotic versus laparoscopic colectomy.

DETAILED DESCRIPTION:
The short-term advantages of minimally invasive colon resection have been well established in several randomized trials. A major factor in the development of morbidity is the surgical stress response with subsequent increased demand on the patient's reserves and immune competence. Although the advantage in term of stress response of laparoscopic surgery over open surgery has been widely reported, little is known about the role of robotic surgery.

Robotic approaches have seen significant growth in the last 5 years. Taking advantage of three-dimensional visualization, improved articulation, and multiple operating arms provides theoretical advantages in colorectal cancer surgery. In an attempt to evaluate the surgical stress response and immune function after robotic colorectal surgery a comparative study has been designed. Two surgical procedures were evaluated: Robotic colorectal resection (Experimental group) and Laparoscopic colorectal resection (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be those with a histologically confirmed malignancy planned for an elective, segmental, curative colectomy

Exclusion Criteria:

* Patients with a previous midline laparotomy, emergency surgery, or immune depressant disease or medication will be excluded from this study. Peri-operative or post-operative complications will be considered exclusion criteria.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
interleukin 1 | change between time before surgery, 24 hours after surgery, 72 hours after surgery
interleukin 6 | change between time before surgery, 24 hours after surgery, 72 hours after surgery
Tumor necrosis factor alpha | change between time before surgery, 24 hours after surgery, 72 hours after surgery
C-reactive protein | change between time before surgery, 24 hours after surgery, 72 hours after surgery
fibrinogen | change between time before surgery, 24 hours after surgery, 72 hours after surgery
prolactin | change between time before surgery, 24 hours after surgery, 72 hours after surgery
cortisol | change between time before surgery, 24 hours after surgery, 72 hours after surgery
insulin | change between time before surgery, 24 hours after surgery, 72 hours after surgery
glucagon | change between time before surgery, 24 hours after surgery, 72 hours after surgery
Adrenocorticotropic hormone | change between time before surgery, 24 hours after surgery, 72 hours after surgery
Growth hormone | change between time before surgery, 24 hours after surgery, 72 hours after surgery
human leukocyte antigen | change between time before surgery, 24 hours after surgery, 72 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided